CLINICAL TRIAL: NCT06068218
Title: Translational Assessment of Vitiligo According to Body Locations Translational Study
Brief Title: Translational Assessment of Vitiligo According to Body Locations
Acronym: Vitiligo BL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23-PP-06
Record Dates: First submitted 2023-09-05; First posted 2023-10-05 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient Group (Other)
  Interventions: Other: Biopsy for the patient group
- Volunteer group (Other)
  Interventions: Other: biopsy for the volunteer group

INTERVENTIONS:
Other: Biopsy for the patient group — The investigator will perform a 4mm skin biopsy will be performed on 5 body sites: neck, trunk, elbows, wrist and feet. For vitiligo patients, the biopsies will be taken on a non-depigmented skin.
  Arms: Patient Group
Other: biopsy for the volunteer group — A publicity in the hospital will announce the study, and will be use to recruit the healthy volunteers. The investigator will perform a 4mm skin biopsy will be performed on 5 body sites: neck, trunk, elbows, wrist and feet.
  Arms: Volunteer group

SUMMARY:
Vitiligo affects 0.5 to 2% of worldwide population and has a demonstrated impact on the quality of life.

Optimal treatment of vitiligo requires to target the auto-immune inflammatory response (to halt the depigmentation process), but also to induce the differentiation of melanocyte stem cells (to induce repigmentation). There is a well demonstrated discrepancy in the repigmentation response between anatomical areas of the body. Face and neck are the best responder with complete or almost complete repigmentation achieved in most cases under treatment. Trunk and limbs could have a complete or almost complete repigmentation in approximately half of the cases. The repigmentation is much more difficult in wrists, elbows, knees, proximal part of the hands. Finally, some areas such as the extremities of hands and feet, palms, soles, are almost impossible to repigment.

The investigator hypothesize that there are some factors that are produced in the skin that prevent (or at least decrease) the differentiation but also probably the migration and proliferation of melanocytes.

Primary objective To compare the mRNA expression of each types of cells in the skin of vitiligo patients compared to healthy volunteers according to body locations

ELIGIBILITY:
Inclusion Criteria:

* Men and women with non-segmental vitiligo for the vitiligo group and men and women without any auto-immune disorder for the control group
* ≥ 18 and <70 years
* For women of child-bearing age, a urine pregnancy test (βHCG in urines) will be performed.
* Affiliation to a social security system
* Signed informed consent

Exclusion Criteria:

* Pregnant women
* Segmental or mixed vitiligo
* Vitiligo with less than 2 years duration
* Skin auto-immune or inflammatory skin disorders other than vitiligo (ie. active atopic dermatitis, psoriasis, lichen planus…)
* Exposure to sun (with intent to tan or repigment the skin) or artificial UV (UV cabins, lamps or lasers) during the month before inclusion
* Concomitant use of topical or systemic immunosuppressive medication or steroids
* Contra-indication to xylocaine with 2 % adrenalin
* Pregnant or breast-feeding women
* Vulnerable people: minors, adult under guardianship or deprived of freedom, adult under curatorship
* Participants in other clinical therapeutic studies involving a drug that could interfere with the present evaluation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-06-18 (Actual); Primary Completion 2026-02-11 (Estimated); Study Completion 2026-04-02 (Estimated)

PRIMARY OUTCOMES:
skin samples | at inclusion
  Transcriptomic profiling by sequencing method will be performed on the skin samples

CONTACTS AND LOCATIONS:
Overall Officials: Passeron Thierry, PhD, Principal Investigator — CHU de Nice, Service de Dermatologie
Locations (1):
- CHU de Nice - Hôpital de l'Archet, Nice, Alpes-maritimes, France

IPD SHARING:
Plan to Share IPD: No